CLINICAL TRIAL: NCT06684145
Title: The Effect Of Kinesiotape Application On Clinical Parameters In Postmenopausal Women With Chronic Low Back Pain: A Randomized Controlled Study
Brief Title: The Effect Of Kinesiotape Application In Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Muhammet Sahin Elbasti, Head of Physiotherapy and Rehabilitation Department, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 163
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Chronic Low-back Pain (cLBP)
Keywords: Chronic low back pain; Kinesiotape; Sleep quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotape application (Experimental): Kinesiotape application will be performed by a certified researcher using 5cm x 5cm kinesiotape material. In addition to the kinesiotape application, patients will be given a 30-day home exercise program. This consists of passive lumbar flexion (single and double leg stretching), hamstring stretching, pelvic tilt, half sit-up, bridge, straight leg raises, and hip and back extensor strengthening exercises.
  Interventions: Other: Kinesiotape application
- Control group (Other): Exercise program will be performed to the control group
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Kinesiotape application — Kinesiotape application will be performed by a certified researcher using 5cm x 5cm kinesiotape material. The standing patient, prepared in terms of clothing and skin, will be asked to lean forward. While adhering the tape to the right paravertebral region, the lower end of the tape will be adhered 7 cm below the sacroiliac joint at the level of the paravertebral muscles. The patient, still leaning forward, will be then asked to make a slight rotation to the left; in this position, the tape will be adhered upwards on the paravertebral muscles without any tension. For the left paravertebral region, the procedure will be reversed as compared to the right, ensuring that the tape was not stretched at all.
  Arms: Kinesiotape application
Other: Exercise — Patients will be given a 30-day home exercise program. This consists of passive lumbar flexion (single and double leg stretching), hamstring stretching, pelvic tilt, half sit-up, bridge, straight leg raises, and hip and back extensor strengthening exercises.
  Arms: Control group

SUMMARY:
This study was conducted to determine the effects of kinesiotaping (KT) and sham KT applied with exercise program on clinical parameters such as pain, sleep, and quality of life in postmenopausal women with chronic low back pain. A randomized controlled experimental design, characteristic of quantitative research, was utilized. The subjects consisted of 60 postmenopausal women. The Visual Analog Scale (VAS), Roland Morris Disability Questionnaire (RMDQ) and Pittsburgh Sleep Quality Index (PSQI) were used as data collection tools.

DETAILED DESCRIPTION:
With rising life expectancy, women are expected to spend a third of their lives in the postmenopausal stage. Consequently, focusing research on postmenopausal women is considered crucial. This study was conducted to determine the effects of kinesiotaping (KT) and sham KT applied with exercise program on clinical parameters such as pain, sleep, and quality of life in postmenopausal women with chronic low back pain. A randomized controlled experimental design, characteristic of quantitative research, was utilized. The subjects consisted of 60 postmenopausal women. The Visual Analog Scale (VAS), Roland Morris Disability Questionnaire (RMDQ) and Pittsburgh Sleep Quality Index (PSQI) were used as data collection tools.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal patients with chronic nonspecific mechanical low back pain for at least three months
* VAS score of at least 3

Exclusion Criteria:

* Patients with a neurologic deficit, history of lumbar surgery, inflammatory low back pain, spinal stenosis, spondylolisthesis, a history of cardiopulmonary disease preventing exercise, severe osteoporosis, or a skin infection in the application area

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-03-10 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | up to 48 hours
  VAS is used to subjectively measure perceived pain. It is a scale in the form of a 0-10 cm ruler, with 'no pain' at one end and 'the most severe pain' at the other, used to quantify pain intensity. The patient marks their pain level on the ruler.

SECONDARY OUTCOMES:
Pittsburgh sleep quality index | up to 48 hours
  Turkish reliability and validity study conducted by Ağargün et al. (1996) this scale, which assesses an individual's sleep quality over the past month, includes 24 items. Of these, 19 are self-reported questions answered by the individual, and five are answered by the roommate or spouse

CONTACTS AND LOCATIONS:
Locations (1):
- Muhammet Şahin Elbastı, Elâzığ, Elâzığ, Turkey (Türkiye)